CLINICAL TRIAL: NCT03273205
Title: The Changes in the Body-perception and Perception of the Pain in Patients With Anorexia Nervosa Before and After Using the tDCS
Brief Title: Transcranial Direct Current Stimulation (tDCS) in the Treatment of Anorexia Nervosa
Acronym: SANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silvie Ceresnakova (Other)
Responsible Party: Sponsor-Investigator, Silvie Ceresnakova, Principal Investigator, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1955/16 S-IV
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Anorexia Nervosa
Keywords: Transcranial direct current stimulation (tDCS)
MeSH Terms: conditions — Anorexia Nervosa | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS (Experimental): The first group of patients has the real stimulation and the electrodes are placed in this position:
  Anode: Left DLPFC [F3) Cathode: Right Supraorbital (FP2)
  Interventions: Device: Anodal tDCS
- Sham tDCS (Sham Comparator): The second group has the sham stimulation, but the electrodes are placed in the same position as in the first group:
  Anode: Left DLPFC [F3) Cathode: Right Supraorbital (FP2)
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Anodal tDCS — This group gets a real stimulation
  Arms: Anodal tDCS
Device: Sham tDCS — This group gets a sham stimulation
  Arms: Sham tDCS

SUMMARY:
Anorexia Nervosa (AN) is a serious and often chronical eating disorder characterized by an extreme effort for weight loss and intense fear of becoming fat despite the obvious thinness. The treatment is very difficult and not always effective. That´s the reason why we are looking for new ways of the therapeutic approach.

Transcranial direct current stimulation (tDCS) is a neuromodulation technique, which modulates the neuronal excitability. According to previous research it has a potential to help people with Anorexia Nervosa.

The device for the tDCS has two electrodes, an anode (the excitatory one) and a cathode (the inhibitory one). We put them on the skull into the different positions, in dependence on the fact, if we want to excite or on to inhibit the parts of the brain under the electrodes.

There are several hypothesis how could the tDCS help in patients with AN. One of them speaks about the hyperactivity of the right hemisphere in Anorexia Nervosa. Therefore could the anodal (excitatory) tDCS over the left hemisphere and the cathodal (inhibitory one) help in resetting the inter-hemispheric balance.

DETAILED DESCRIPTION:
Stimulation of 2 milliampere is applied for 30 minutes in every real session. Together there are 10 sessions, the application is every workday within 2 weeks.

All measurements and questionnaires are made 4 times:

1. Before the stimulation
2. On the day of the last stimulation
3. 14 days after the last stimulation
4. 28 days after the last stimulation

ELIGIBILITY:
Inclusion Criteria:

* patients with the diagnosis of anorexia nervosa

Exclusion Criteria:

* patients: with the diagnosis of epilepsy, after a serious injury of head, with chronic headache, with some metal or electronic implants in their heads and patients who are pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change of the Eating Disorders Examination Questionnaire (EDEq) score | 8 weeks
  Comparison of the total scores and subscores of the Eating Disorders Examination Questionnaire (EDEq)

SECONDARY OUTCOMES:
Change of the Zung Self-Rating Depression Scale | 8 weeks
  Comparison of the total scores of the Zung Self-Rating Depression Scale
Change of the pain threshold | 8 weeks
  Measurement of the pain threshold with the TSA II Neuro Sensory Analyzer
Change of the weight in kilograms | 8 weeks
  Regularly weighting on the scale

CONTACTS AND LOCATIONS:
Overall Officials: Hana Papezova, Prof.,M.D.,CSc., Study Director — Department of Psychiatry, Charles University in Prague and General University Hospital in Prague
Locations (1):
- Department of Psychiatry, Charles University in Prague and General University Hospital in Prague, Prague, Czechia

REFERENCES:
- [Derived] Baumann S, Mares T, Albrecht J, Anders M, Vochoskova K, Hill M, Bulant J, Yamamotova A, Stastny O, Novak T, Holanova P, Lambertova A, Papezova H. Effects of Transcranial Direct Current Stimulation Treatment for Anorexia Nervosa. Front Psychiatry. 2021 Oct 6;12:717255. doi: 10.3389/fpsyt.2021.717255. eCollection 2021. PMID 34690831